CLINICAL TRIAL: NCT02779699
Title: Phase I Study of Tolerance and Pharmacokinetics of AL2846 in Patients With Advanced Cancer
Brief Title: A Study of AL2846 on Tolerance and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL2846-I-0001
Record Dates: First submitted 2016-05-16; First posted 2016-05-20 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL2846 (Experimental): AL2846 QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: AL2846

INTERVENTIONS:
Drug: AL2846 — AL2846 p.o. qd

SUMMARY:
A study of AL2846,a C-met/Hepatocyte growth factor tyrosine kinase inhibitor,in patients with advanced cancer.

DETAILED DESCRIPTION:
To study the pharmacokinetic characteristics of AL2846 in the human body; To recommend a reasonable dose and indication for subsequent research.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of Advanced solid tumors（especially Hepatocellular Carcinoma and Lung Cancer ）,at least one measurable lesion (by RECIST1.1)
* Lack of the standard treatment or treatment failure
* 18-65 years,ECOG PS:0-1,Life expectancy of more than 3 months
* 30 Days or more from the last cytotoxic therapy
* Main organs function is normal
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped
* Patients should participate in the study voluntarily and sign informed consent

Exclusion Criteria:

* Patients suffering from other malignancies currently or ever, except for cured cervical carcinoma in situ, non-melanoma skin cancers
* Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea, intestinal obstruction etc.)
* Patients participated in other anticancer drug clinical trials within 4 weeks or Patients participating in other clinical trials now
* Blood pressure unable to be controlled ideally by one drug(systolic pressure≥140 mmHg，diastolic pressure≥90 mmHg); Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias(including male QTc≥450ms,female QTc≥470ms) and patients with Grade 1 or higher congestive heart failure (NYHA Classification)
* Urine protein ≥ ++，and 24-hour urinary protein excretion>1.0 g confirmed
* Patients with non-healing wounds or fractures
* Patients with drug abuse history and unable to get rid of or Patients with mental disorders
* History of immunodeficiency
* Patients with concomitant diseases which could seriously endanger their own safety or could affect completion of the study according to investigators' judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The type of dose-limiting toxicity(ies) (DLT[s]) of AL2846 | For 4 weeks for DLTs
  Subjects within 28 days after treatment appear the following toxicity reaction relate to the drug ：II °or above of kidney damage，III °or above of non-hematological toxicity,IV°hematological toxicity ,Neutropenia associated with fever.
Pharmacokinetics of AL2846 (in plasma) | up to 28 Days (endpoint when the two consecutive time points of blood drug concentration <150 DPM/mL)
  In the study of single-dose, full PK profiles will be obtained at H0/H0.5/H1/H2/H4/H8/H11/H24/H34/H48/H58/H72/H96/H120/H168 (H means Hour). In the study of multiple-dose, full PK profiles will be obtained at D0/D1/D4/D7/D10/D13/D15/D18/D21/D24/D28 (D means Day).
The maximum tolerated dose (MTD) of AL2846 | 48 weeks
  The highest dose at which no more than 33% of the subjects experience a dose-limiting toxicity (DLT) during treatment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 56 days up to intolerance the toxicity or PD (up to 24 months)
  Percentage of participants with OR based assessment of confirmed complete remission (CR) or confirmed partial remission (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided